CLINICAL TRIAL: NCT04404699
Title: Stimulation Testing Performed During TcPO2 Measurement Improve the Diagnosis of Peripheral Arterial Disease in Patients With Diabetic Foot: A Multicentre Trial
Brief Title: Stimulation TcPO2 Test in the PAD Diagnosis in Diabetic Foot
Acronym: stimTcPO2
Status: Completed | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: General University Hospital, Prague (Other); Motol University Hospital (Other)
Responsible Party: Principal Investigator, Vladimíra Fejfarová, Principal investigator, Institute for Clinical and Experimental Medicine
Other Study IDs: TcPO2SDN
Record Dates: First submitted 2020-05-09; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Peripheral Arterial Disease
Keywords: diabetic foot; peripheral arterial disease; TcPO2
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stimulation TcPO2 test — During measurement of TcPO2 in various angiosomes the stimulation test will be performed. We modify the Ratschow test (elevation of the lower limbs, rhythmic flexion and extension in talocrural joints for 2 minutes, then return to horizontal position). TcPO2 is measured continuously. Depending on the type of detected flows by DUS in the evaluated arteries supplying the relevant angiosome, in which TcPO2 values are measured, the patients and their angiosomes will be divided into 2 baseline groups - group M with monophasic flows or arterial obliterations and group T with triphasic flows.
  We will compare macrocirculation parameters-systolic pressure on dorsalis pedis artery (DPA), posterior tibial artery (PTA) and their doppler indexes. The resting TcPO2, the minimal TcPO2 found during the stimulation test, their delta (resting TcPO2 - minimal TcPO2) and the percentage decrease in TcPO2 will be compared between the study groups, as well as the duration of TcPO2 recovery.

SUMMARY:
All diagnostic procedures of peripheral arterial disease (PAD) in the diabetic foot (DF) are limited due to diabetes mellitus and its late complications. The aim of our study is to refine the diagnosis of peripheral arterial disease (PAD) by a new transcutaneous oximetry (TcPO2) stimulation test (a modified Ratschow test) in patients with diabetic foot.

DETAILED DESCRIPTION:
Patients with diabetic foot and mild to moderate PAD (WIfI - Ischemia 1 or 2) with baseline TcPO2 values 30-50 mmHg will be included into the study. TcPO2 will be measured on the feet in different angiosomes. During this measurement a stimulation test consisting of a modified Ratschow test involving 2 minutes of exercise will be conducted. Specific TcPO2 parameters will be assessed during the whole procedure (resting TcPO2 before stimulation test, minimal TcPO2, delta TcPO2 (minimum TcPo2 minus resting TcPO2) percentage decrease of TcPO2 during the stimulation test and TcPO2 recovery time (time to the adjustment of TcPO2 to the resting values).

All TcPO2 parameters detected during TcPO2 stimulation test will be correlated with parameters of macrocirculation (systolic blood pressures (SBP) on tibial arteries and their Ankle-Brachial Indexes (ABI), toe pressures (TP) and toe-brachial indexesTBI) and DUS findings (monophasic/triphasic flow in relevant artery supplying measured angiosome)

ELIGIBILITY:
Inclusion Criteria:

* presence of Diabetic Foot in patients with type 1 or type 2 diabetes mellitus, with WIfI classification of ischemia 1-2 (based on TcPO2) without previously diagnosed PAD or with known PAD based on the patients' history or previous vascular reconstruction (endovascular or surgical vascular interventions)
* resting TcPO2 values between 30-50 mm Hg.

Exclusion Criteria:

* vascular interventions on evaluated limb within 12 months prior to the enrolment into the study
* factors possibly influencing for example oxygen saturation or feet movement:

  * patient imobility
  * impairment of movements at the talocrural joints
  * vasculitis
  * heart failure or advanced COPD
  * severe anaemia (plasma haemoglobin below 8g / dL)
  * hypoperfusion due to shock or cardiac dysfunction
  * sepsis
  * massive swelling of the lower limbs of various ethiology (including lymphedema)
  * active Charcot osteoarthropathy
  * critical limb ischemia with WIfI classification of ischemia 3
  * lower limb claudication below 200m
  * venous insufficiency of CEAP classification 6
  * severe diabetic kidney disease (CKD stage 4 or 5)

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with diabetic foot treated in out-patient foot clinic predominantly for diabetic foot ulcers
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in TcPO2 | 30 minutes
  How change special parameters evaluated during Stimulation TcPO2 test
Correlation of stimulation TcPO2 parameters with the type of peripheral arterial flow | 30 minutes
  A correlation of special parameters detected during Stimulation TcPO2 test with the type of arterial flow in large vessels supplying measured angiosome by TcPO2 will be performed

SECONDARY OUTCOMES:
Correlation of stimulation TcPO2 parameters with macrocirculation parameters | 30 minutes
  A correlation of special parameters detected during Stimulation TcPO2 test with the large vessels parameters usually used for PAD diagnosis (systolic blood pressures on ADP, PTA and their ABI and toe pressures and their TBI

CONTACTS AND LOCATIONS:
Locations (1):
- IKEM, Prague, Czechia

REFERENCES:
- [Derived] Fejfarova V, Matuska J, Jude E, Pithova P, Flekac M, Roztocil K, Woskova V, Dubsky M, Jirkovska A, Bem R, Husakova J, Lanska V. Stimulation TcPO2 Testing Improves Diagnosis of Peripheral Arterial Disease in Patients With Diabetic Foot. Front Endocrinol (Lausanne). 2021 Dec 10;12:744195. doi: 10.3389/fendo.2021.744195. eCollection 2021. PMID 34956078